CLINICAL TRIAL: NCT05525000
Title: Validity and Reliability of Consumer-Grade Optical Heart Rate Sensors to Assess Volume of Physical Activity and to Categorize Its Intensity
Brief Title: Validity and Reliability of Optical Heart Rate Sensors
Acronym: ValOpti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Collaborators: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Mahdi Sareban, Priv.-Doz. Dr. Dr. med., Salzburger Landeskliniken
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ValOpti
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Validation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants aged over 35 (Experimental): Participants run through our validation protocol
  Interventions: Device: Validation

INTERVENTIONS:
Device: Validation — The validation protocol consists of the following activities:
  Activities of daily living, Exercise test on the treadmill, Exercise test on the cycle ergometer, Free-living session

SUMMARY:
To evaluate validity and reliability of consumer-grade optical heart-rate devices we aim to compare these devices with medical-grade ECG. The design includes an extended and practical validation protocol for consumer-grade optical heart rate devices in laboratory and ambulatory free-living conditions using a medical-grade ECG device as a criterion measure.

DETAILED DESCRIPTION:
Candidate consumer-grade wearables are selected according to available data from manufacturers, available scientific literature and our team's own practical experience.

First, a mobile 12-lead ECG (Amedtec ECGpro, Aue, Germany) device is placed on the participant according to recommendations of medical societies and the manufacturer's instructions. Additionally, the participant wears four optical heart rate devices simultaneously. Each device will be placed according to the manufacturer's instructions, The devices will be randomly applied on the dominant or non-dominant wrist and to the dominant and non-dominant arm, respectively. All participants will be handed an instruction sheet and video how to place each device in case it is displaced and how to check that data collection is working.

The 13-min laboratory protocol will be performed in keeping with an expert statement of the INTERLIVE Network and starts with a session mimicking lifestyle activity that consists of: 1 minute of quiet sitting, 2 minutes of upper body activities, 1 minute of quiet sitting, 30 seconds of transition to treadmill, 2 minutes of walking at self-selected speed, 30 seconds of transition to chair, 2 minutes of seated typing, 30 seconds of transition, 2 minutes of full body daily living activities including vacuum cleaning and ironing, and 1 minute of quiet sitting.

After completion of the lifestyle activities test, participants proceed with the treadmill step test. The treadmill step test protocol starts with 1 minute of quiet standing, 3 minutes of (4 km/h), 30 seconds of rest, 3 minutes of running (6 km/h) and an increment of 2 km/h at each stage with 30 seconds of rest between each stage until volitional exhaustion. Capillary blood samples will be taken from the earlobe to assess blood lactate concentration after each stage of the exercise test. Dependent on physical fitness 3 to 8 blood lactate samples will be taken. A breath-by-breath spiroergometry device will measure gas exchange, ventilation and maximal oxygen uptake during the exercise test using a metabolic analyzer. After termination of the exercise test subjective exhaustion will be assessed by the BORG scale. The 12-lead ECG will allow ruling out clinically relevant coronary artery disease and/or arrhythmias, and identify maximum heart rates from which intensity zones will be derived. Test termination will be followed by a 5-min cool down period at walking speed (3 km/h) on the treadmill. Throughout the treadmill test the participant is secured with a safety belt to prevent any injuries in case of falling.

Directly after the 5-min cool down, exercise testing on the cycle ergometer starts, beginning with 1 minute of quiet sitting. Then load is increased until the participant exercises at low intensity (57-63% of maximum heart rate obtained in the treadmill test) which will be maintained for at least 2 minutes, followed by 1 minute of rest, 2 minutes of moderate intensity (64-76% of maximum heart rate), 1 minute of rest, 2 minutes of vigorous intensity (>77% of maximum heart rate) followed by 1 minute of cool-down. All activity intensity zones are defined according to medical guidelines.

For the free-living part the electrodes of an ambulatory 3-lead-ECG (Amedtec ECGpro, Aue, Germany) are placed according to the manufacturer's instructions. Additionally, the participant wears four optical heart rate devices simultaneously.

The measurement of all devices starts simultaneously between 8:00 and 11:00 a.m. and is recorded for 24 hours. The only instruction the participants get are to walk for six minutes on a flat terrain as fast as possible once in the afternoon. At the end of the 24-hour period, participants stop all optical heart rate devices and return the devices to the University Institute of Sports Medicine, Prevention and Rehabilitation. There, the lifestyle activities and cycle ergometry laboratory testing protocol of day 1 will be repeated for reliability assessment. Finally, participants will be asked to fill out the IDEA-Fast Technology Experience Questionnaire (ITEQ) questionnaire to obtain information on the usability of the devices.

The 3-lead Holter-ECG will be analyzed by a licensed cardiologist for relevant arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 80 years
* All sexes
* Able to perform physical activity according to the study protocol
* Written informed consent

Exclusion Criteria:

* Acute infections and/or diseases
* Diseases limiting walking distance and/or physical activity outlined in the study protocol
* Atrial fibrillation
* Clinical signs of chronic venous insufficiency ≥ 1 at upper extremities
* Obesity WHO grade 2 or more (Body Mass Index >35 kg/m²)
* Skin wound or tattoo where wearables are placed
* Pregnancy

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 24 hours
  Heart rate is measured with different devices and ECG while performing different activities and free living

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsinstitut für präventive und rehabilitative Sportmedizin, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neudorfer M, Kumar D, Smeddinck JD, Kulnik ST, Niebauer J, Treff G, Sareban M. Validity of Four Consumer-Grade Optical Heart Rate Sensors for Assessing Volume and Intensity Distribution of Physical Activity. Scand J Med Sci Sports. 2024 Nov;34(11):e14756. doi: 10.1111/sms.14756. PMID 39508366